CLINICAL TRIAL: NCT06783465
Title: AI-Driven Generative Content and Precision Dynamic Executive Function Cognitive Digital Therapeutics System for Dementia Management
Brief Title: AI-Driven Cognitive Digital Therapeutics for Dementia Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202404013
Record Dates: First submitted 2024-09-15; First posted 2025-01-20 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Digital therapeutics session three times per week
  Interventions: Device: Digital therapeutics session
- Control (No Intervention)

INTERVENTIONS:
Device: Digital therapeutics session — During the digital therapeutics session, the patient performs tasks by handling objects according to instructions displayed by the device. A camera records the task performance, and the system analyzes the task performance.
  Arms: Intervention

SUMMARY:
The study would investigate the effect of a cognitive digital therapeutics system. The intervention group would receive three digital therapeutics sessions per week for 8 weeks, while the control group would receive usual care. Evaluations would be done at baseline, week 8, and week 16.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 50 years old.
2. Clinical Dementia Rating from 0.5-1
3. Physician diagnosed mild neurocognitive disorder or dementia (according to ICD-11 diagnostic criteria)

Exclusion Criteria:

1. Mini-mental state examination score below 18
2. If receiving an approved Alzheimer's disease treatment such as acetylcholinesterase inhibitor (AChEIs) or memantine or both for Alzheimer's disease, must be on a stable dose for at least 4 weeks prior to Baseline.
3. Any neurological condition that may be contributing to cognitive impairment above and beyond that caused by the participant's mild neurocognitive disorder or dementia.
4. History of transient ischemic attacks (TIA), stroke, or seizures within 12 months of Screening.
5. Any psychiatric diagnosis or symptoms (example, hallucinations, major depression, or delusions) that could interfere with study procedures in the participant.
6. Geriatric Depression Scale (GDS) score greater than or equal to 10 at Screening.
7. Participants who were dosed in a clinical study involving any new chemical entities for AD within 6 months prior to screening unless it can be documented that the participant was in a placebo treatment arm.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Instrumental Activities of Daily Living (IADL) | Baseline, Week 8, Week 16
  e.g., K-IADL (Korean Instrumental Activities of Daily Living): range from 0 to 33; Higher scores = worse outcomes, lower scores = better independence.

SECONDARY OUTCOMES:
The Montreal Cognitive Assessment (MoCA) | Baseline, Week 8, Week 16
  Range: 0 to 30; Higher scores indicate better cognitive function.
Mini-Mental State Examination score (MMSE) | Baseline, Week 8, Week 16
  Range: 0 to 30; Higher scores indicate better cognitive function.
Clinical Dementia Rating score (CDR) | Baseline, Week 8, Week 16
  Range: 0 to 3; Higher scores indicate greater severity of dementia.
Executive Function Performance Test score (EFPT) | Baseline, Week 8, Week 16
  Range: 0 to 100; Higher scores indicate worse executive functioning.

OTHER OUTCOMES:
Geriatric Depression Scale (GDS-15) | Baseline, Week 8, Week 16
  Range: 0 to 15; Higher scores indicate greater levels of depressive symptoms.
The Family Confusion Assessment Method (FAM-CAM) | Baseline, Week 8, Week 16
  Range: Scored as present or absent; Presence indicates delirium.
Activities of Daily Living (ADL) score | Baseline, Week 8, Week 16
  Higher scores indicate greater independence: e.g., Katz ADL--range from 0 to 6; Barthel Index--range from 0 to 100.
WAIS-III Digit span forward, backward, and sequencing | Baseline, Week 8, Week 16
  Range: Variable (raw scores depend on the total number of correct trials, typically ranging from 0 to ~30, depending on individual performance).
  Standardized Scoring: Raw scores are converted to age-specific scaled scores, typically ranging from 1 to 19.
  Interpretation: Higher scores indicate better short-term memory, working memory, and cognitive processing capacity.
Frontal assessment battery (FAB) subtest 5 | Baseline, Week 8, Week 16
  Range: 0 to 3. Interpretation: Higher scores indicate better motor programming and cognitive flexibility, reflecting improved frontal lobe function.
Zarit Burden Interview (ZBI) | Baseline, Week 8, Week 16
  Range: 0 to 88 (for the full scale) Interpretation: Higher scores indicate greater caregiver burden.
Neuropsychiatric Inventory (NPI) | Baseline, Week 8, Week 16
  Range: 0 to 144; Higher scores indicate more severe neuropsychiatric symptoms across assessed domains
Quality of Life Outcome for Patients with Neurologic Conditions (PROMIS) | Baseline, Week 8, Week 16
  Range: Standardized T-score, typically 20 to 80; Higher scores can indicate better or worse outcomes depending on the specific domain

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Wan Fang Hospital, Taipei City, Taipei, Taiwan